CLINICAL TRIAL: NCT03709797
Title: Effectiveness of Dry Needling as a Treatment of Shoulder Myofascial Pain Syndrome in Spinal Cord Injury Patients: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Dry Needling as a Treatment of Shoulder Myofascial Pain Syndrome in Spinal Cord Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Sandra Palacios Alfonso, PhD Student, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULeon-020-2018
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Spinal Cord Injuries; Myofascial Pain Syndrome; Shoulder Pain; Puncture
Keywords: Spinal Cord Injury; Shoulder Pain; Myofascial Pain Syndrome; Dry Needling
MeSH Terms: conditions — Spinal Cord Injuries; Myofascial Pain Syndromes; Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will receive dry needling treatment.
  Interventions: Procedure: Dry needling in infraspinatus muscle
- Control group (Sham Comparator): Control group will receive sham dry needling treatment.
  Interventions: Procedure: Dry needling in infraspinatus muscle

INTERVENTIONS:
Procedure: Dry needling in infraspinatus muscle — Dry needling technique with multiple rapid needle insertion.

SUMMARY:
Shoulder pain in people with spinal cord injury is one of the most prevalent in acute and chronic patients because of weakness in shoulder periarticular muscles, and also because of overuse of these part of the body in assistive devices.

This study aims to evidence if dry needling (a physiotherapy technique) is also useful in patients with spinal cord injury, and how long it could hold out without or less pain.

ELIGIBILITY:
Inclusion Criteria:

* At least one year after Spinal Cord Injury (chronic patients).
* Spinal Cord Injury under C5-C6 spinal level with American Spinal Injury Association (ASIA) classification.
* Patients with shoulder pain and at least one active trigger point in infraspinatus muscle.

Exclusion Criteria:

* Be apprehensive to the needles (belonephobia).
* Immunosuppression.
* Drug instability.
* Other medical causes that, under medical prescription, dry needling in the shoulder are discouraged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand Spanish version (DASHe). | Change from baseline and one week later.
  In upper limb pathology this test evaluates functional activities in relation to the difficulty involved in performing them with a score between 1 and 5.
  The DASHe questionnaire consists of a main part of 30 items, and two specific modules for people who work with musical instruments / sports or for the workplace. In this study, only the main part has been used. The 30 items have a score of 1 to 5, with 5 being the maximum of the valued symptom, and at least 27 questions of 3 must be answered.
  The disability / symptom score will therefore be between 0 (best possible score) and 100 (worst possible score).

SECONDARY OUTCOMES:
Pressure Pain Thershold (algometry). | Change from baseline, immediately after intervention and one week later.
  Baseline®dolorimeter - 22lb / 10kg, STOCK CODE: 12-1442 It will be measured with an algometer that is an instrument that provides quantitative / objective information on pain at a specific point, depending on the pressure on which it is applied. A circle is drawn around the trigger point on which the indelible marker test will be performed to confirm in the last measurement which is the exact point on which it is worked. 3 consecutive measurements are made at the same point, waiting between one and another measurement for a period between 30-60 seconds, and the average of the 3 measurements will be used as a statistical value.
McGill Pain Questionnaire (Spanish version). | Change from baseline and one week later.
  This scale consists of a set of 78 adjectives included in 20 groups (including 2 to 6 in each group) and that express a characteristic of pain. Within these 20 groups we find the Pain Rating Index (PRI) divided into: sensory (groups 1-10), affective (groups 11-15), evaluative (group 16) and miscellaneous (group 17-20) ), of which the patient can only choose one word from each of the 20 groups, choosing only those adjectives that best suit his pain sensation. It also includes a category on the changes that experimental pain, and another with a rate of pain intensity (Present Pain Index = PPI).
Visual Analog Scale (VAS) | Change from baseline and one week later.
  This scale is a line of 10 centimeters without marks between the parameters without pain and unbearable pain, where the patient has to mark between those parameters where his pain is.
Shoulder Pain And Disability Index Spanish version (SPADIe). | Change from baseline and one week later.
  It consists of a 10-item scale that assesses shoulder pain and the difficulties in activities of daily life that it generates, divided into two main sections: the first 4 items refer to the intensity of pain and the last 6 refer to the difficulty of carrying out specific activities. All the items have a minimum score of 0 and a maximum of 10, therefore the total score is between 0 and 100, with 0 being the best possible value in relation to pain and difficulty, and 100 being the highest value and so much more painful and disabling.
Range Of Movement (ROM) | Change from baseline, immediately after intervention and one week later.
  Objective will be to measure different ranges of movement of the affected upper limb (internal rotation and horizontal adduction) in question due to myofascial pain syndrome. In this case the movements that passively will be measured with a bubble inclinometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Palacios Alfonso, Burgos, Spain